CLINICAL TRIAL: NCT02928406
Title: An Open Label, Single Arm, Multicenter, Safety Study of Atezolizumab in Locally Advanced or Metastatic Urothelial or Non-Urothelial Carcinoma of the Urinary Tract
Brief Title: A Study of Atezolizumab in Locally Advanced or Metastatic Urothelial or Non-Urothelial Carcinoma of the Urinary Tract
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO29983; 2016-002625-11 (EudraCT Number)
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Urinary Tract Cancer
MeSH Terms: conditions — Urologic Neoplasms | interventions — atezolizumab

ARMS (1):
- Atezolizumab (Experimental): Participants will receive atezolizumab every 3 weeks (Q3W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 milligrams (mg) will be administered by intravenous (IV) infusion Q3W.
  Other Names: MPDL3280A

SUMMARY:
This Phase IIIb, multicenter study will assess the safety of atezolizumab as second- to fourth-line treatment for participants with locally advanced or metastatic urothelial or non-urothelial cancer of the urinary tract in addition to evaluate the efficacy of atezolizumab and potential tumor biomarkers associated with atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically documented locally advanced (tumor [T] 4b, any node [N]; or any T, N 2-3) or metastatic (M1, Stage IV) urothelial or non-urothelial carcinoma of the urinary tract
* Participants with measurable and/or non-measurable disease according to RECIST v1.1
* Participants must have progressed during or following treatment with at least one prior (and not more than 3) treatments for inoperable, locally advanced or metastatic urothelial or non-urothelial carcinoma of the urinary tract
* If available, a representative formalin-fixed paraffin-embedded (FFPE) tumor specimen block should be submitted
* Eastern cooperative oncology group (ECOG) performance status 0, 1 or 2

Exclusion Criteria:

* Treatment with more than three prior lines of systemic therapy for inoperable, locally advanced or metastatic urothelial or non-urothelial carcinoma of the urinary tract
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to study treatment initiation

  1. Participants who were in another clinical trial with therapeutic intent within 4 weeks of study treatment initiation but were not on active drug in that prior trial are eligible
  2. Participants who were in another clinical trial with therapeutic intent within 4 weeks of study treatment initiation but were in the follow-up phase of that prior trial and had stopped receiving active drug 4 or more weeks before study treatment initiation are eligible
* Malignancies other than the one studied in this protocol within 5 years prior to Cycle 1, Day 1
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol
* Significant renal disorder indicating a need for renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (175):
- Argentina (3):
  - Inst. Alexander Fleming; Oncologia, Buenos Aires
  - Hospital Aleman, Caba
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
- Australia (10):
  - Canberra Hospital; Medical Oncology, Canberra, Australian Capital Territory
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Prince of Wales Hospital; Oncology, Randwick, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital; Hematology/Oncology, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Hospital Olivia Newton John Cancer Centre, Heidelberg, Victoria
- Austria (5):
  - Medizinische Universität Innsbruck; Universitätsklinik für Urologie, Innsbruck
  - Ordensklinikum Linz Elisabethinen; Abteilung für Urologie und Andrologie, Linz
  - Landeskrankenhaus Salzburg; Universitätsklinik für Urologie und Andrologie der PMU, Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
  - Medizinische Universität Wien; Universitätsklinik für Urologie, Vienna
- Belgium (4):
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
- Brazil (6):
  - Pronutrir - suporte nutricional e quimioterapia ltda., Fortaleza, Ceará
  - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- Bulgaria (3):
  - Complex Oncology Center (COC)-Plovidiv, Plovdiv
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - SHATOD - Sofia, Sofia
- Canada (5):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Ontario
  - The Ottawa Hospital Cancer Center; General Campus, Ottawa, Ontario
- Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, China
- Clinica del Country, Bogotá, Colombia
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni Thomayerova Nemocnice; Onkologicke Oddeleni, Prague
- Denmark (4):
  - Aalborg Universitetshospital; Onkologisk Afdeling, Aalborg
  - Aarhus Universitetshospital; Kræftafdelingen, Aarhus N
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Rigshospitalet; Onkologisk Klinik, København Ø
- Estonia (2):
  - East Tallinn Central Hospital; Clinic of Internal Medicine, Tallinn
  - North Estonia Medical Centre Foundation; Oncology Center, Tallinn
- Germany (12):
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Urologie, Dresden
  - Universitätsklinikum Erlangen; Medizinische Klinik 5 - Hämatound Internist Onko, Erlangen
  - Universitätsmedizin Göttingen Georg-August-Universität; Klinik für Urologie, Göttingen
  - Krankenhaus Martha-Maria Halle-Dölau, Klinik für Urologie, Halle
  - Medizinische Hochschule Hannover; Klinik für Urologie und Onkologische Urologie, Hanover
  - Onkologische Schwerpunktpraxis, Heidelberg
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Urologie, Lübeck
  - Kliniken Maria Hilf GmbH, Krankenhaus St. Franziskus, Mönchengladbach
  - Klinikum rechts der Isar der TU München; Urologische Klinik und Poliklinik, München
  - Universitätsklinikum Münster, Klinik für Urologie und Kinderurologie, Münster
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
  - Universitätsklinikum Ulm; Klinik für Urologie, Ulm
- Greece (7):
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - IASO General Hospital of Athens, Athens
  - Agioi Anargyroi Cancer Hospital; 2Nd Oncology Dept., Kifissia
  - Metropolitan Hospital; 2Nd Oncology Clinic, Piraeus
  - Thermi Clinic; Oncology Clinic, Thermi Thessalonikis
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Hungary (5):
  - Honvédelmi Minisztérium Állami Egészségügyi Központ; Onkológiai Osztály; Oncology department, Budapest
  - Semmelwies University of Medicine; Urology Dept., Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház; Onkológiai Osztály, Szolnok
- India (4):
  - HealthCare Global Cancer Centre; Medical Oncology, Ahmedabad, Gujarat
  - Artemis Health Institute, Gurgaon, Haryana
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - TATA Medical Centre; Medical Oncology, Kolkata, West Bengal
- Ireland (2):
  - Cork University Hospital, Cork
  - Adelaide & Meath Hospital, Dublin, Incorporating the National Children's Hospital; Oncology Day Unit, Dublin
- Italy (26):
  - Policlinico Ospedaliero Ss Annunziata; U.O. Di Clinica Oncologica, Chieti, Abruzzo
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - ISTITUTO NAZIONALE TUMORI IRCCS FONDAZIONE G. PASCALE; Dipartimento Uro-Ginecologico, Napoli, Campania
  - AZ.Osp S. Orsola ? Malpighi-Reparto di Oncologia Medica, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Oncologia, Reggio Emilia, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia, Udine, Friuli Venezia Giulia
  - Policlinico Universitario Campus Biomedico Di Roma; U.O.Oncologia Medica, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini; Oncologia Medica, Rome, Lazio
  - Policlinico Universitario "Agostino Gemelli"; U.O.C. Oncologia Medica, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - ASST DI CREMONA; Dip. Medicina - S.C. Oncologia, Cremona, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - A.O. UNIVERSITARIA S. LUIGI GONZAGA; Oncologia Medica, Orbassano, Piedmont
  - A.O.U. Cagliari-P.O. Monserrato;U.O. Oncologia, Cagliari, Sardinia
  - Ospedale Cannizzaro, Oncologia, Catania, Sicily
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato;U.O.C. Oncologia, Arezzo, Tuscany
  - Azlenda Ospendaliero-Universitaria Pisana; C.O. Oncologia 2, Pisa, Tuscany
  - Azienda Ospedaliera S. Maria - Terni; Oncologia, Terni, Umbria
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Prima, Padua, Veneto
  - Azienda Ospedaliera di Verona-Policlinico G.B. Rossi; Oncologia Medica, Verona, Veneto
- Hotel Dieu de France; Oncology, Beirut, Lebanon
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics - Endocrinology clinic, Kaunas
  - National Cancer Institute, Vilnius
- Netherlands (5):
  - NKI/AvL, Amsterdam
  - VU MEDISCH CENTRUM; Dept. of Medical Oncology, Amsterdam
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Maastricht University Medical Centre; Medical Oncology, Maastricht
  - St. Antonius locatie Leidsche Rijn, Utrecht
- Poland (4):
  - NZOZ Onko-Dent G. L. Slomian, Spolka Jawna, ?ory
  - Centrum Onkologii Ziemi LUBELSKIEJ im. Sw Jana z Dukli, I oddz. Chemioterapii, Lublin
  - Szpital Kliniczny Przemienienia Pa?skiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Szpital Grochowski im. dr med. Rafa?a Masztaka Sp. z o.o., Warsaw
- Portugal (4):
  - Hospital de Braga; Servico de Oncologia Medica X, Braga
  - HUC; Servico de Urologia e Transplantacao Renal, Coimbra
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Romania (5):
  - Oncopremium Team Srl, Baia Mare
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca; Spital de zi-Parter, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Centrul de Radioterapie AMETHYST, Floreşti
  - Oncomed SRL; Oncologie, Timișoara
- Russia (2):
  - Blokhin Cancer Research Center; Urological Dept, Moscow, Moscow Oblast
  - P.A. Herzen Oncological Inst. ; Oncology, Moscow, Moscow Oblast
- King Faisal Specialist Hospital & Research Centre; Oncology, Riyadh, Saudi Arabia
- Narodny onkologicky ustav, Bratislava, Slovakia
- Spain (32):
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Complejo Hospitalario de Althaia; Servicio de Oncologia, Manresa, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital de Basurto; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital del Mar Barcelona, Barcelona
  - Hospital Clínic i Provincial; Servicio de Oncología, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Oncologia, Girona
  - Hospital General Universitario de Guadalajara; Servicio de Oncologia, Guadalajara
  - Hospital Lucus Augusti; Servicio de Oncologia, Lugo
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Oncologia, Murcia
  - Complejo Hospitalario de Orense; Servicio de Oncologia, Ourense
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Oncologia, Toledo
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Hospital La Fe, Valencia
- Switzerland (7):
  - Universitaetsspital Basel; Onkologie, Basel
  - Ospedale Regionale di Bellinzona Medizin Onkologie, Bellinzona
  - Inselspital Bern; Universitätsklinik für Medizinische Onkologie, Klinische Forschungseinheit, Bern
  - Kantonsspital Graubünden Medizin Onkologie; Onkologie und Hämatologie, Chur
  - Hôpitaux Universit. de Genève Médecine Oncologie; Oncologie, Geneva
  - Luzerner Kantonsspital; Medizinische Onkologie, Lucerne
  - Kantonsspital Winterthur; Medizinische Onkologie, Winterthur
- Taiwan (2):
  - National Cheng Kung Uni Hospital; Dept of Hematology and Oncology, Tainan
  - Chang Gung Medical Foundation-Linkou, Urinary Oncology, Taoyuan District
- United Kingdom (5):
  - Velindre Cancer Centre, Cardiff
  - Raigmore Hospital; Dept of Radiotherapy & Oncology, Inverness
  - Leicester Royal Infirmary NHS Trust, Leicester
  - Barts and the London NHS Trust., London
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Bamias A, Merseburger A, Loriot Y, James N, Choy E, Castellano D, Lopez-Rios F, Calabro F, Kramer M, de Velasco G, Zakopoulou R, Tzannis K, Sternberg CN. New prognostic model in patients with advanced urothelial carcinoma treated with second-line immune checkpoint inhibitors. J Immunother Cancer. 2023 Jan;11(1):e005977. doi: 10.1136/jitc-2022-005977. PMID 36627145
- [Derived] Bamias A, Merseburger AS, Loriot Y, James N, Choy E, Castellano D, Lopez-Rios F, Calabro F, Kramer M, de Velasco G, Zakopoulou R, Tzannis K, Sternberg CN. SAUL, a single-arm study of atezolizumab for chemotherapy-pretreated locally advanced or metastatic carcinoma of the urinary tract: outcomes by key baseline factors, PD-L1 expression and prior platinum therapy. ESMO Open. 2021 Jun;6(3):100152. doi: 10.1016/j.esmoop.2021.100152. Epub 2021 May 10. PMID 33984672
- [Derived] Merseburger AS, Castellano D, Powles T, Loriot Y, Retz M, Voortman J, Huddart RA, Gedye C, Van Der Heijden MS, Gurney H, Ong M, de Ducla S, Pavlova J, Fear S, Sternberg CN. Safety and Efficacy of Atezolizumab in Understudied Populations with Pretreated Urinary Tract Carcinoma: Subgroup Analyses of the SAUL Study in Real-World Practice. J Urol. 2021 Aug;206(2):240-251. doi: 10.1097/JU.0000000000001768. Epub 2021 Apr 9. PMID 33835866
- [Derived] Loriot Y, Sternberg CN, Castellano D, Oosting SF, Dumez H, Huddart R, Vianna K, Alonso Gordoa T, Skoneczna I, Fay AP, Nole F, Massari F, Brasiuniene B, Maroto P, Fear S, Di Nucci F, de Ducla S, Choy E. Safety and efficacy of atezolizumab in patients with autoimmune disease: Subgroup analysis of the SAUL study in locally advanced/metastatic urinary tract carcinoma. Eur J Cancer. 2020 Oct;138:202-211. doi: 10.1016/j.ejca.2020.07.023. Epub 2020 Sep 6. PMID 32905959
- [Derived] Cathomas R, Schardt J, Pless M, Llado A, Mach N, Riklin C, Haefeli J, Fear S, Stenner F. Swiss experience of atezolizumab for platinum-pretreated urinary tract carcinoma: the SAUL study in real-world practice. Swiss Med Wkly. 2020 May 4;150:w20223. doi: 10.4414/smw.2020.20223. eCollection 2020 May 4. PMID 32399958
- [Derived] Sternberg CN, Loriot Y, James N, Choy E, Castellano D, Lopez-Rios F, Banna GL, De Giorgi U, Masini C, Bamias A, Garcia Del Muro X, Duran I, Powles T, Gamulin M, Zengerling F, Geczi L, Gedye C, de Ducla S, Fear S, Merseburger AS. Primary Results from SAUL, a Multinational Single-arm Safety Study of Atezolizumab Therapy for Locally Advanced or Metastatic Urothelial or Nonurothelial Carcinoma of the Urinary Tract. Eur Urol. 2019 Jul;76(1):73-81. doi: 10.1016/j.eururo.2019.03.015. Epub 2019 Mar 23. PMID 30910346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 172 centers in 32 countries
Groups:
- Atezolizumab: Participants received atezolizumab every 3 weeks (Q3W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurred first).
Period: Overall Study
Arm/Group | Atezolizumab
Started | 1004
Did Not Receive Study Drug | 7
Completed | 0
Not Completed | 1004
Not completed — Death | 780
Not completed — Progressive disease | 3
Not completed — Lost to Follow-up | 49
Not completed — Non-compliance | 2
Not completed — Withdrawal by Subject | 40
Not completed — Study terminated by sponsor | 57
Not completed — Physician Decision | 1
Not completed — Various reasons | 72

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who had received at least 1 dose of atezolizumab. The safety population was used for all baseline and safety analyses.
Arm/Group | Atezolizumab
Number analyzed (Participants) | 997
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (10.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225
  Male | 772
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 112
  Not Hispanic or Latino | 820
  Unknown or Not Reported | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 920
  More than one race | 0
  Unknown or Not Reported | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: AEs were defined as any untoward medical occurrence in a subject administered a pharmaceutical product, regardless of causal attribution. An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. New disease, exacerbation of existing disease, recurrence of an intermittent medical condition not present at baseline, any deterioration in a laboratory value or other clinical test associated with symptoms or leading to a change in study/concomitant treatment or discontinuation from study drug as well as events related to protocol-mandated interventions are considered AEs.
Time Frame: Baseline up to end of study (up to approximately 6 years)
Population: The safety population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 997
Participants | 900

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as date of death (due to any cause) or censoring minus date of start of study treatment plus 1.
Time Frame: Randomization until death from any cause (up to approximately 6 years)
Population: The intent-to-treat (ITT) population included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 1004
Months | 8.57 [7.75 to 9.72]

3. Secondary Outcome: Progression Free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS was defined as the date of first occurrence of tumor progression (earliest of the dates of the RECIST component indicating tumor progression) or date of death (in the absence of tumor progression) by any cause, whichever occurred first, or date of censoring minus date of start of study treatment plus 1.
Time Frame: Randomization up to disease progression or death from any cause, whichever occurred first (up to approximately 6 years)
Population: The ITT population included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 1004
Months | 2.20 [2.14 to 2.40]

4. Secondary Outcome: PFS as Per Modified Response Evaluation Criteria in Solid Tumors (Modified RECIST)
Description: PFS as per Modified RECIST was defined as:
  * date of first occurrence of tumor progression after a modified confirmed response if the participant was a responder according to modified RECIST or
  * date of first occurrence of tumor progression in case the participant was not a responder according to modified RECIST or
  * date of death (in the absence of tumor progression) by any cause, or
  * date of censoring whichever occurred first, minus date of start of study treatment plus 1
Time Frame: Randomization up to disease progression or death from any cause, whichever occurred first (up to approximately 6 years)
Population: The ITT population included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 1004
Months | 2.79 [2.37 to 3.45]

5. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) as Assessed by RECIST v1.1
Description: BOR was assessed by the investigators according to the RECIST v1.1. BOR was defined as a complete response (CR) or partial response (PR) determined on two consecutive investigator assessments >= 4 weeks apart in participants with measurable disease at baseline. CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 millimeters (mm); PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must have demonstrated an absolute increase of at least 5 mm. Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: Randomization up to disease progression or death from any cause, whichever occurred first (up to approximately 6 years)
Population: The ITT population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 1004
Percentage of participants | 15.7 [13.5 to 18.1]

6. Secondary Outcome: Percentage of Participants With BOR as Assessed by Modified RECIST
Description: BOR was assessed by the investigators according to the modified RECIST. BOR was defined as complete response (CR) or partial response (PR). CR includes complete disappearance of all tumor lesions and no new measurable or unmeasurable lesions confirmed by a consecutive assessment >=4 weeks from the first documented date. PR is a decrease in the sum of the diameters of all target and all new measurable lesions >=30%, relative to baseline, in the absence of CR confirmed by a consecutive assessment >=4 weeks from the first documented date. The assessment of BOR included post-screening RECIST assessments obtained up to: 1) death from any cause, 2) last evaluable RECIST assessment in the absence of death, 3) start of a subsequent anti-cancer therapy, whichever occurred first.
Time Frame: Randomization up to disease progression or death from any cause, whichever occurred first (up to approximately 6 years)
Population: The ITT population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 1004
Percentage of participants | 16.4 [14.2 to 18.9]

7. Secondary Outcome: Percentage of Participants With Disease Control as Assessed by RECIST v1.1
Description: Disease control was determined separately on disease status using RECIST v1.1 by the investigator. Disease control rate was defined as the sum of the complete response, partial response, and stable disease rates.
Time Frame: Randomization up to disease progression or death from any cause, whichever occurred first (up to approximately 6 years)
Population: The ITT population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 1004
Percentage of participants | 39.9 [36.9 to 43.0]

8. Secondary Outcome: Percentage of Participants With Disease Control as Assessed by Modified RECIST
Description: Disease control was determined separately on disease status using modified RECIST by the investigator. Disease control rate was defined as the sum of the complete response, partial response, and stable disease rates.
Time Frame: Randomization up to disease progression or death from any cause, whichever occurred first (up to approximately 6 years)
Population: The ITT population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 1004
Percentage of participants | 46.0 [42.9 to 49.2]

9. Secondary Outcome: Duration of Response (DOR) as Assessed by RECIST v1.1
Description: Duration of response was determined separately on disease status using RECIST v1.1 by the investigator. For overall responders, DoR was defined as the time from the date of first occurrence of a confirmed response (complete response or partial response) to date of tumor progression or death from any cause, or to censoring date: 1) end of response coincided with the date of tumor progression or death (in the absence of tumor progression) used for the PFS endpoint, 2) for a participant without disease progression or death following a response, the censored end of response coincided with the PFS censoring date (that was latest RECIST assessment or start of subsequent cancer therapy, whichever occurred first).
Time Frame: Time from first occurrence of a documented response to disease progression or death from any cause, whichever occurred first (up to approximately 6 years)
Population: The ITT population included all enrolled participants. Only participants with a response were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 158
Months | 27.79 [18.89 to 43.30]

10. Secondary Outcome: DOR as Assessed by Modified RECIST
Description: Duration of response was determined separately on disease status using modified RECIST by the investigator. For overall responders, DoR was defined as the time from the date of first occurrence of a confirmed response (complete response or partial response) to date of tumor progression following that confirmed response or death from any cause, or to censoring date: 1) end of response was the date of tumor progression after that confirmed response or death (in the absence of tumor progression), 2) for a participant without disease progression or death following a response, the censored end of response was the latest RECIST assessment or start of subsequent cancer therapy, whichever occurred first.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 165
Months | 29.73 [21.72 to 43.30]

11. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL), as Assessed Using European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) Score
Description: The EORTC QLQ-C30 included global health status, functional scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea/vomiting, and pain) and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Most questions used a 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores were averaged and transformed to 0 - 100 scale. Higher scores on the global health status and functional scales indicated better health status/function. Higher scores on the symptoms scales and symptom items indicated greater symptom burden.
Time Frame: Baseline, Day 1 of Cycles 1, 2, 3 and thereafter every 9 weeks for 54 weeks from study treatment start; and then every 12 weeks until progression/study discontinuation (up to approximately 6 years) (Cycle length = 21 days)
Population: The ITT population included all enrolled participants who completed the questionnaire at baseline and had 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Atezolizumab
Number analyzed (Participants) | 964
Score on a scale
  Physical score Baseline: number analyzed (Participants) | 963
  Physical score Baseline | 70.62 (23.784)
  Physical score Cycle(C) 2 Day(D) 1: number analyzed (Participants) | 812
  Physical score Cycle(C) 2 Day(D) 1 | -3.43 (16.923)
  Physical score C3D1: number analyzed (Participants) | 710
  Physical score C3D1 | -3.98 (18.854)
  Physical score C4D1: number analyzed (Participants) | 526
  Physical score C4D1 | -2.01 (18.647)
  Physical score C7D1: number analyzed (Participants) | 345
  Physical score C7D1 | 1.72 (19.408)
  Physical score C10D1: number analyzed (Participants) | 275
  Physical score C10D1 | 3.10 (17.494)
  Physical score C13D1: number analyzed (Participants) | 223
  Physical score C13D1 | 3.32 (16.829)
  Physical score C16D1: number analyzed (Participants) | 187
  Physical score C16D1 | 3.62 (19.790)
  Physical score C19D1: number analyzed (Participants) | 159
  Physical score C19D1 | 3.27 (20.591)
  Physical score C23D1: number analyzed (Participants) | 129
  Physical score C23D1 | 4.16 (19.298)
  Physical score C27D1: number analyzed (Participants) | 121
  Physical score C27D1 | 4.90 (20.032)
  Physical score C31D1: number analyzed (Participants) | 108
  Physical score C31D1 | 6.50 (20.053)
  Physical score C35D1: number analyzed (Participants) | 102
  Physical score C35D1 | 4.95 (24.876)
  Physical score C39D1: number analyzed (Participants) | 91
  Physical score C39D1 | 7.33 (22.307)
  Physical score C43D1: number analyzed (Participants) | 76
  Physical score C43D1 | 6.06 (19.840)
  Physical score C47D1: number analyzed (Participants) | 74
  Physical score C47D1 | 6.56 (19.682)
  Physical score C51D1: number analyzed (Participants) | 70
  Physical score C51D1 | 4.85 (22.585)
  Physical score C55D1: number analyzed (Participants) | 55
  Physical score C55D1 | 4.93 (19.110)
  Physical score C59D1: number analyzed (Participants) | 54
  Physical score C59D1 | 5.68 (21.916)
  Physical score C63D1: number analyzed (Participants) | 53
  Physical score C63D1 | 7.64 (18.894)
  Physical score C67D1: number analyzed (Participants) | 46
  Physical score C67D1 | 8.66 (23.154)
  Physical score C71D1: number analyzed (Participants) | 42
  Physical score C71D1 | 3.50 (19.652)
  Physical score C75D1: number analyzed (Participants) | 24
  Physical score C75D1 | 6.67 (17.914)
  Physical score C79D1: number analyzed (Participants) | 20
  Physical score C79D1 | 1.00 (18.245)
  Physical score C83D1: number analyzed (Participants) | 8
  Physical score C83D1 | -4.15 (7.908)
  Physical score C87D1: number analyzed (Participants) | 2
  Physical score C87D1 | -10.00 (14.142)
  Physical score C91D1: number analyzed (Participants) | 1
  Physical score C91D1 | -20.00
  Physical score Discontinuation visit: number analyzed (Participants) | 443
  Physical score Discontinuation visit | -13.87 (26.541)
  Role score Baseline: number analyzed (Participants) | 962
  Role score Baseline | 67.29 (31.545)
  Role score C2D1: number analyzed (Participants) | 814
  Role score C2D1 | -5.38 (25.918)
  Role score C3D1: number analyzed (Participants) | 712
  Role score C3D1 | -4.31 (27.800)
  Role score C4D1: number analyzed (Participants) | 529
  Role score C4D1 | -1.45 (29.012)
  Role score C7D1: number analyzed (Participants) | 351
  Role score C7D1 | 1.81 (29.762)
  Role score C10D1: number analyzed (Participants) | 277
  Role score C10D1 | 3.25 (27.060)
  Role score C13D1: number analyzed (Participants) | 224
  Role score C13D1 | 5.73 (26.659)
  Role score C16D1: number analyzed (Participants) | 187
  Role score C16D1 | 4.10 (28.314)
  Role score C19D1: number analyzed (Participants) | 161
  Role score C19D1 | 2.28 (28.107)
  Role score C23D1: number analyzed (Participants) | 130
  Role score C23D1 | 2.70 (32.535)
  Role score C27D1: number analyzed (Participants) | 122
  Role score C27D1 | 6.56 (30.725)
  Role score C31D1: number analyzed (Participants) | 109
  Role score C31D1 | 9.18 (31.951)
  Role score C35D1: number analyzed (Participants) | 103
  Role score C35D1 | 4.86 (34.899)
  Role score C39D1: number analyzed (Participants) | 91
  Role score C39D1 | 10.81 (33.457)
  Role score C43D1: number analyzed (Participants) | 76
  Role score C43D1 | 6.58 (31.276)
  Role score C47D1: number analyzed (Participants) | 74
  Role score C47D1 | 7.21 (31.464)
  Role score C51D1: number analyzed (Participants) | 70
  Role score C51D1 | 6.91 (31.914)
  Role score C55D1: number analyzed (Participants) | 56
  Role score C55D1 | 5.06 (27.136)
  Role score C59D1: number analyzed (Participants) | 54
  Role score C59D1 | 8.03 (23.736)
  Role score C63D1: number analyzed (Participants) | 53
  Role score C63D1 | 5.66 (24.664)
  Role score C67D1: number analyzed (Participants) | 46
  Role score C67D1 | 2.90 (34.116)
  Role score C71D1: number analyzed (Participants) | 43
  Role score C71D1 | 4.65 (29.171)
  Role score C75D1: number analyzed (Participants) | 24
  Role score C75D1 | 5.57 (22.335)
  Role score C79D1: number analyzed (Participants) | 20
  Role score C79D1 | 4.18 (31.934)
  Role score C83D1: number analyzed (Participants) | 8
  Role score C83D1 | -4.16 (14.743)
  Role score C87D1: number analyzed (Participants) | 2
  Role score C87D1 | -8.30 (11.738)
  Role score C91D1: number analyzed (Participants) | 1
  Role score C91D1 | -16.60
  Role score Discontinuation visit: number analyzed (Participants) | 443
  Role score Discontinuation visit | -17.61 (35.664)
  Emotional score Baseline: number analyzed (Participants) | 961
  Emotional score Baseline | 75.89 (22.274)
  Emotional score C2D1: number analyzed (Participants) | 809
  Emotional score C2D1 | 0.79 (18.975)
  Emotional score C3D1: number analyzed (Participants) | 706
  Emotional score C3D1 | 1.55 (18.868)
  Emotional score C4D1: number analyzed (Participants) | 525
  Emotional score C4D1 | 1.04 (19.530)
  Emotional score C7D1: number analyzed (Participants) | 348
  Emotional score C7D1 | 3.05 (18.978)
  Emotional score C10D1: number analyzed (Participants) | 278
  Emotional score C10D1 | 4.39 (17.733)
  Emotional score C13D1: number analyzed (Participants) | 222
  Emotional score C13D1 | 3.96 (17.669)
  Emotional score C16D1: number analyzed (Participants) | 188
  Emotional score C16D1 | 5.79 (20.044)
  Emotional score C19D1: number analyzed (Participants) | 161
  Emotional score C19D1 | 4.90 (20.156)
  Emotional score C23D1: number analyzed (Participants) | 130
  Emotional score C23D1 | 5.45 (20.057)
  Emotional score C27D1: number analyzed (Participants) | 122
  Emotional score C27D1 | 5.94 (19.538)
  Emotional score C31D1: number analyzed (Participants) | 109
  Emotional score C31D1 | 10.17 (19.057)
  Emotional score C35D1: number analyzed (Participants) | 103
  Emotional score C35D1 | 8.90 (19.361)
  Emotional score C39D1: number analyzed (Participants) | 91
  Emotional score C39D1 | 9.80 (20.883)
  Emotional score C43D1: number analyzed (Participants) | 76
  Emotional score C43D1 | 8.22 (20.618)
  Emotional score C47D1: number analyzed (Participants) | 74
  Emotional score C47D1 | 7.21 (19.762)
  Emotional score C51D1: number analyzed (Participants) | 71
  Emotional score C51D1 | 9.23 (20.377)
  Emotional score C55D1: number analyzed (Participants) | 56
  Emotional score C55D1 | 8.48 (18.359)
  Emotional score C59D1: number analyzed (Participants) | 54
  Emotional score C59D1 | 9.88 (17.890)
  Emotional score C63D1: number analyzed (Participants) | 53
  Emotional score C63D1 | 9.12 (16.766)
  Emotional score C67D1: number analyzed (Participants) | 46
  Emotional score C67D1 | 8.52 (20.452)
  Emotional score C71D1: number analyzed (Participants) | 43
  Emotional score C71D1 | 7.56 (18.345)
  Emotional score C75D1: number analyzed (Participants) | 25
  Emotional score C75D1 | 7.33 (21.430)
  Emotional score C79D1: number analyzed (Participants) | 20
  Emotional score C79D1 | 5.84 (22.465)
  Emotional score C83D1: number analyzed (Participants) | 8
  Emotional score C83D1 | 8.34 (8.913)
  Emotional score C87D1: number analyzed (Participants) | 2
  Emotional score C87D1 | 0.00 (47.235)
  Emotional score C91D1: number analyzed (Participants) | 1
  Emotional score C91D1 | -33.40
  Emotional score Discontinuation visit: number analyzed (Participants) | 442
  Emotional score Discontinuation visit | -7.49 (23.771)
  Cognitive score Baseline: number analyzed (Participants) | 962
  Cognitive score Baseline | 85.43 (20.943)
  Cognitive score C2D1: number analyzed (Participants) | 811
  Cognitive score C2D1 | -1.83 (19.255)
  Cognitive score C3D1: number analyzed (Participants) | 707
  Cognitive score C3D1 | -2.40 (18.344)
  Cognitive score C4D1: number analyzed (Participants) | 526
  Cognitive score C4D1 | -1.58 (15.886)
  Cognitive score C7D1: number analyzed (Participants) | 348
  Cognitive score C7D1 | 0.00 (16.737)
  Cognitive score C10D1: number analyzed (Participants) | 278
  Cognitive score C10D1 | -0.78 (16.763)
  Cognitive score C13D1: number analyzed (Participants) | 222
  Cognitive score C13D1 | -0.37 (14.476)
  Cognitive score C16D1: number analyzed (Participants) | 188
  Cognitive score C16D1 | 0.44 (16.743)
  Cognitive score C19D1: number analyzed (Participants) | 161
  Cognitive score C19D1 | -0.10 (17.221)
  Cognitive score C23D1: number analyzed (Participants) | 131
  Cognitive score C23D1 | -1.27 (17.973)
  Cognitive score C27D1: number analyzed (Participants) | 122
  Cognitive score C27D1 | -0.68 (17.324)
  Cognitive score C31D1: number analyzed (Participants) | 109
  Cognitive score C31D1 | 1.38 (14.715)
  Cognitive score C35D1: number analyzed (Participants) | 103
  Cognitive score C35D1 | 0.32 (15.112)
  Cognitive score C39D1: number analyzed (Participants) | 91
  Cognitive score C39D1 | -1.46 (15.238)
  Cognitive score C43D1: number analyzed (Participants) | 76
  Cognitive score C43D1 | -2.19 (16.623)
  Cognitive score C47D1: number analyzed (Participants) | 74
  Cognitive score C47D1 | -0.68 (14.702)
  Cognitive score C51D1: number analyzed (Participants) | 71
  Cognitive score C51D1 | -0.23 (16.051)
  Cognitive score C55D1: number analyzed (Participants) | 56
  Cognitive score C55D1 | 1.79 (14.791)
  Cognitive score C59D1: number analyzed (Participants) | 54
  Cognitive score C59D1 | -0.31 (17.271)
  Cognitive score C63D1: number analyzed (Participants) | 53
  Cognitive score C63D1 | -1.25 (15.615)
  Cognitive score C67D1: number analyzed (Participants) | 46
  Cognitive score C67D1 | -3.98 (16.909)
  Cognitive score C71D1: number analyzed (Participants) | 43
  Cognitive score C71D1 | -5.42 (13.946)
  Cognitive score C75D1: number analyzed (Participants) | 25
  Cognitive score C75D1 | -6.67 (15.951)
  Cognitive score C79D1: number analyzed (Participants) | 20
  Cognitive score C79D1 | -8.34 (13.792)
  Cognitive score C83D1: number analyzed (Participants) | 8
  Cognitive score C83D1 | -6.24 (12.382)
  Cognitive score C87D1: number analyzed (Participants) | 2
  Cognitive score C87D1 | 0.00 (0.00)
  Cognitive score C91D1: number analyzed (Participants) | 1
  Cognitive score C91D1 | 0.00
  Cognitive score Discontinuation visit: number analyzed (Participants) | 444
  Cognitive score Discontinuation visit | -9.76 (23.884)
  Social score Baseline: number analyzed (Participants) | 961
  Social score Baseline | 74.56 (26.597)
  Social score C2D1: number analyzed (Participants) | 813
  Social score C2D1 | -1.25 (26.277)
  Social score C3D1: number analyzed (Participants) | 705
  Social score C3D1 | -0.02 (24.058)
  Social score C4D1: number analyzed (Participants) | 526
  Social score C4D1 | -0.38 (25.568)
  Social score C7D1: number analyzed (Participants) | 347
  Social score C7D1 | 0.24 (26.865)
  Social score C10D1: number analyzed (Participants) | 278
  Social score C10D1 | 3.78 (25.930)
  Social score C13D1: number analyzed (Participants) | 222
  Social score C13D1 | 4.43 (23.550)
  Social score C16D1: number analyzed (Participants) | 188
  Social score C16D1 | 3.99 (23.579)
  Social score C19D1: number analyzed (Participants) | 161
  Social score C19D1 | 4.45 (25.186)
  Social score C23D1: number analyzed (Participants) | 131
  Social score C23D1 | 1.65 (28.106)
  Social score C27D1: number analyzed (Participants) | 122
  Social score C27D1 | 4.24 (24.482)
  Social score C31D1: number analyzed (Participants) | 109
  Social score C31D1 | 7.65 (28.007)
  Social score C35D1: number analyzed (Participants) | 103
  Social score C35D1 | 5.02 (26.279)
  Social score C39D1: number analyzed (Participants) | 91
  Social score C39D1 | 6.96 (26.070)
  Social score C43D1: number analyzed (Participants) | 76
  Social score C43D1 | 5.26 (25.704)
  Social score C47D1: number analyzed (Participants) | 74
  Social score C47D1 | 4.96 (27.412)
  Social score C51D1: number analyzed (Participants) | 71
  Social score C51D1 | 6.34 (24.541)
  Social score C55D1: number analyzed (Participants) | 56
  Social score C55D1 | 6.55 (21.946)
  Social score C59D1: number analyzed (Participants) | 54
  Social score C59D1 | 8.03 (22.369)
  Social score C63D1: number analyzed (Participants) | 53
  Social score C63D1 | 6.29 (22.695)
  Social score C67D1: number analyzed (Participants) | 46
  Social score C67D1 | 5.80 (27.491)
  Social score C71D1: number analyzed (Participants) | 43
  Social score C71D1 | 3.50 (21.995)
  Social score C75D1: number analyzed (Participants) | 25
  Social score C75D1 | 10.01 (22.041)
  Social score C79D1: number analyzed (Participants) | 20
  Social score C79D1 | 5.84 (28.767)
  Social score C83D1: number analyzed (Participants) | 8
  Social score C83D1 | 18.75 (27.383)
  Social score C87D1: number analyzed (Participants) | 2
  Social score C87D1 | 8.30 (11.738)
  Social score C91D1: number analyzed (Participants) | 1
  Social score C91D1 | 33.30
  Social score Discontinuation visit: number analyzed (Participants) | 444
  Social score Discontinuation visit | -12.20 (33.586)
  Fatigue score Baseline: number analyzed (Participants) | 963
  Fatigue score Baseline | 36.04 (26.343)
  Fatigue score C2D1: number analyzed (Participants) | 814
  Fatigue score C2D1 | 5.58 (22.444)
  Fatigue score C3D1: number analyzed (Participants) | 712
  Fatigue score C3D1 | 5.01 (23.869)
  Fatigue score C4D1: number analyzed (Participants) | 528
  Fatigue score C4D1 | 3.27 (23.637)
  Fatigue score C7D1: number analyzed (Participants) | 349
  Fatigue score C7D1 | -2.56 (24.879)
  Fatigue score C10D1: number analyzed (Participants) | 277
  Fatigue score C10D1 | -3.95 (23.633)
  Fatigue score C13D1: number analyzed (Participants) | 224
  Fatigue score C13D1 | -2.46 (23.492)
  Fatigue score C16D1: number analyzed (Participants) | 189
  Fatigue score C16D1 | -4.97 (25.081)
  Fatigue score C19D1: number analyzed (Participants) | 161
  Fatigue score C19D1 | -4.73 (26.358)
  Fatigue score C23D1: number analyzed (Participants) | 130
  Fatigue score C23D1 | -3.34 (26.603)
  Fatigue score C27D1: number analyzed (Participants) | 122
  Fatigue score C27D1 | -6.01 (24.252)
  Fatigue score C31D1: number analyzed (Participants) | 109
  Fatigue score C31D1 | -10.09 (25.731)
  Fatigue score C35D1: number analyzed (Participants) | 103
  Fatigue score C35D1 | -8.95 (28.738)
  Fatigue score C39D1: number analyzed (Participants) | 91
  Fatigue score C39D1 | -9.76 (28.299)
  Fatigue score C43D1: number analyzed (Participants) | 76
  Fatigue score C43D1 | -7.75 (28.295)
  Fatigue score C47D1: number analyzed (Participants) | 74
  Fatigue score C47D1 | -7.95 (24.164)
  Fatigue score C51D1: number analyzed (Participants) | 70
  Fatigue score C51D1 | -9.68 (25.102)
  Fatigue score C55D1: number analyzed (Participants) | 56
  Fatigue score C55D1 | -7.73 (24.710)
  Fatigue score C59D1: number analyzed (Participants) | 54
  Fatigue score C59D1 | -9.46 (21.528)
  Fatigue score C63D1: number analyzed (Participants) | 53
  Fatigue score C63D1 | -7.13 (21.259)
  Fatigue score C67D1: number analyzed (Participants) | 46
  Fatigue score C67D1 | -6.76 (28.838)
  Fatigue score C71D1: number analyzed (Participants) | 43
  Fatigue score C71D1 | -5.42 (23.187)
  Fatigue score C75D1: number analyzed (Participants) | 24
  Fatigue score C75D1 | -3.70 (26.146)
  Fatigue score C79D1: number analyzed (Participants) | 20
  Fatigue score C79D1 | -6.66 (23.200)
  Fatigue score C83D1: number analyzed (Participants) | 8
  Fatigue score C83D1 | -4.18 (13.215)
  Fatigue score C87D1: number analyzed (Participants) | 2
  Fatigue score C87D1 | -5.55 (39.386)
  Fatigue score C91D1: number analyzed (Participants) | 1
  Fatigue score C91D1 | 22.30
  Fatigue score Discontinuation visit: number analyzed (Participants) | 446
  Fatigue score Discontinuation visit | 13.35 (28.962)
  Nausea/Vomiting score Baseline: number analyzed (Participants) | 963
  Nausea/Vomiting score Baseline | 6.94 (14.538)
  Nausea/Vomiting score C2D1: number analyzed (Participants) | 811
  Nausea/Vomiting score C2D1 | 3.53 (16.328)
  Nausea/Vomiting score C3D1: number analyzed (Participants) | 712
  Nausea/Vomiting score C3D1 | 2.43 (15.445)
  Nausea/Vomiting score C4D1: number analyzed (Participants) | 528
  Nausea/Vomiting score C4D1 | 1.77 (14.485)
  Nausea/Vomiting score C7D1: number analyzed (Participants) | 349
  Nausea/Vomiting score C7D1 | 0.81 (14.300)
  Nausea/Vomiting score C10D1: number analyzed (Participants) | 277
  Nausea/Vomiting score C10D1 | -0.36 (12.603)
  Nausea/Vomiting score C13D1: number analyzed (Participants) | 224
  Nausea/Vomiting score C13D1 | -0.52 (11.533)
  Nausea/Vomiting score C16D1: number analyzed (Participants) | 189
  Nausea/Vomiting score C16D1 | -1.06 (12.109)
  Nausea/Vomiting score C19D1: number analyzed (Participants) | 161
  Nausea/Vomiting score C19D1 | -0.72 (10.436)
  Nausea/Vomiting score C23D1: number analyzed (Participants) | 130
  Nausea/Vomiting score C23D1 | 0.13 (10.880)
  Nausea/Vomiting score C27D1: number analyzed (Participants) | 122
  Nausea/Vomiting score C27D1 | -0.14 (11.838)
  Nausea/Vomiting score C31D1: number analyzed (Participants) | 109
  Nausea/Vomiting score C31D1 | -1.53 (8.939)
  Nausea/Vomiting score C35D1: number analyzed (Participants) | 103
  Nausea/Vomiting score C35D1 | -2.91 (9.461)
  Nausea/Vomiting score C39D1: number analyzed (Participants) | 91
  Nausea/Vomiting score C39D1 | -2.93 (10.421)
  Nausea/Vomiting score C43D1: number analyzed (Participants) | 76
  Nausea/Vomiting score C43D1 | -3.29 (8.614)
  Nausea/Vomiting score C47D1: number analyzed (Participants) | 74
  Nausea/Vomiting score C47D1 | -2.93 (8.879)
  Nausea/Vomiting score C51D1: number analyzed (Participants) | 70
  Nausea/Vomiting score C51D1 | -2.86 (8.960)
  Nausea/Vomiting score C55D1: number analyzed (Participants) | 55
  Nausea/Vomiting score C55D1 | -3.03 (9.123)
  Nausea/Vomiting score C59D1: number analyzed (Participants) | 54
  Nausea/Vomiting score C59D1 | -2.47 (9.388)
  Nausea/Vomiting score C63D1: number analyzed (Participants) | 53
  Nausea/Vomiting score C63D1 | -3.46 (9.446)
  Nausea/Vomiting score C67D1: number analyzed (Participants) | 46
  Nausea/Vomiting score C67D1 | -2.90 (9.494)
  Nausea/Vomiting score C71D1: number analyzed (Participants) | 43
  Nausea/Vomiting score C71D1 | -2.33 (8.587)
  Nausea/Vomiting score C75D1: number analyzed (Participants) | 24
  Nausea/Vomiting score C75D1 | -2.09 (5.642)
  Nausea/Vomiting score C79D1: number analyzed (Participants) | 20
  Nausea/Vomiting score C79D1 | -2.51 (6.118)
  Nausea/Vomiting score C83D1: number analyzed (Participants) | 8
  Nausea/Vomiting score C83D1 | 0.00 (0.000)
  Nausea/Vomiting score C87D1: number analyzed (Participants) | 2
  Nausea/Vomiting score C87D1 | 8.30 (11.738)
  Nausea/Vomiting score C91D1: number analyzed (Participants) | 1
  Nausea/Vomiting score C91D1 | 0.00
  Nausea/Vomiting score Discontinuation visit: number analyzed (Participants) | 444
  Nausea/Vomiting score Discontinuation visit | 4.69 (19.358)
  Pain score Baseline | 33.97 (31.221)
  Pain score C2D1: number analyzed (Participants) | 817
  Pain score C2D1 | 0.06 (23.064)
  Pain score C3D1: number analyzed (Participants) | 713
  Pain score C3D1 | 1.54 (26.411)
  Pain score C4D1: number analyzed (Participants) | 529
  Pain score C4D1 | -0.13 (27.312)
  Pain score C7D1: number analyzed (Participants) | 351
  Pain score C7D1 | -2.61 (30.687)
  Pain score C10D1: number analyzed (Participants) | 278
  Pain score C10D1 | -3.90 (26.146)
  Pain score C13D1: number analyzed (Participants) | 224
  Pain score C13D1 | -4.02 (25.814)
  Pain score C16D1: number analyzed (Participants) | 189
  Pain score C16D1 | -5.74 (29.692)
  Pain score C19D1: number analyzed (Participants) | 161
  Pain score C19D1 | -6.83 (27.035)
  Pain score C23D1: number analyzed (Participants) | 131
  Pain score C23D1 | -5.98 (28.577)
  Pain score C27D1: number analyzed (Participants) | 122
  Pain score C27D1 | -9.29 (26.684)
  Pain score C31D1: number analyzed (Participants) | 109
  Pain score C31D1 | -10.10 (25.864)
  Pain score C35D1: number analyzed (Participants) | 103
  Pain score C35D1 | -9.71 (33.050)
  Pain score C39D1: number analyzed (Participants) | 91
  Pain score C39D1 | -11.54 (30.400)
  Pain score C43D1: number analyzed (Participants) | 76
  Pain score C43D1 | -8.56 (29.125)
  Pain score C47D1: number analyzed (Participants) | 74
  Pain score C47D1 | -10.36 (29.157)
  Pain score C51D1: number analyzed (Participants) | 71
  Pain score C51D1 | -6.58 (29.875)
  Pain score C55D1: number analyzed (Participants) | 56
  Pain score C55D1 | -8.04 (26.779)
  Pain score C59D1: number analyzed (Participants) | 54
  Pain score C59D1 | -8.96 (27.033)
  Pain score C63D1: number analyzed (Participants) | 53
  Pain score C63D1 | -5.04 (30.238)
  Pain score C67D1: number analyzed (Participants) | 46
  Pain score C67D1 | -5.80 (32.632)
  Pain score C71D1: number analyzed (Participants) | 43
  Pain score C71D1 | -8.54 (29.178)
  Pain score C75D1: number analyzed (Participants) | 25
  Pain score C75D1 | -12.01 (30.999)
  Pain score C79D1: number analyzed (Participants) | 20
  Pain score C79D1 | -6.67 (32.628)
  Pain score C83D1: number analyzed (Participants) | 8
  Pain score C83D1 | -8.35 (30.876)
  Pain score C87D1: number analyzed (Participants) | 2
  Pain score C87D1 | -16.70 (23.617)
  Pain score C91D1: number analyzed (Participants) | 1
  Pain score C91D1 | 33.30
  Pain score Discontinuation visit: number analyzed (Participants) | 446
  Pain score Discontinuation visit | 9.53 (33.994)
  Dyspnoea score Baseline: number analyzed (Participants) | 961
  Dyspnoea score Baseline | 16.23 (24.815)
  Dyspnoea score C2D1: number analyzed (Participants) | 810
  Dyspnoea score C2D1 | 1.03 (22.912)
  Dyspnoea score C3D1: number analyzed (Participants) | 709
  Dyspnoea score C3D1 | 3.29 (24.647)
  Dyspnoea score C4D1: number analyzed (Participants) | 527
  Dyspnoea score C4D1 | 0.88 (22.962)
  Dyspnoea score C7D1: number analyzed (Participants) | 350
  Dyspnoea score C7D1 | -0.57 (23.661)
  Dyspnoea score C10D1: number analyzed (Participants) | 276
  Dyspnoea score C10D1 | -1.09 (22.079)
  Dyspnoea score C13D1: number analyzed (Participants) | 224
  Dyspnoea score C13D1 | -0.30 (23.616)
  Dyspnoea score C16D1: number analyzed (Participants) | 188
  Dyspnoea score C16D1 | -1.06 (22.042)
  Dyspnoea score C19D1: number analyzed (Participants) | 159
  Dyspnoea score C19D1 | -0.21 (22.650)
  Dyspnoea score C23D1: number analyzed (Participants) | 130
  Dyspnoea score C23D1 | -0.26 (24.014)
  Dyspnoea score C27D1: number analyzed (Participants) | 121
  Dyspnoea score C27D1 | 1.10 (25.791)
  Dyspnoea score C31D1: number analyzed (Participants) | 109
  Dyspnoea score C31D1 | -3.98 (24.725)
  Dyspnoea score C35D1: number analyzed (Participants) | 103
  Dyspnoea score C35D1 | -4.20 (23.647)
  Dyspnoea score C39D1: number analyzed (Participants) | 91
  Dyspnoea score C39D1 | -3.30 (22.794)
  Dyspnoea score C43D1: number analyzed (Participants) | 76
  Dyspnoea score C43D1 | -2.63 (24.798)
  Dyspnoea score C47D1: number analyzed (Participants) | 73
  Dyspnoea score C47D1 | -3.19 (23.669)
  Dyspnoea score C51D1: number analyzed (Participants) | 69
  Dyspnoea score C51D1 | -2.90 (23.379)
  Dyspnoea score C55D1: number analyzed (Participants) | 56
  Dyspnoea score C55D1 | -2.97 (20.366)
  Dyspnoea score C59D1: number analyzed (Participants) | 54
  Dyspnoea score C59D1 | -1.24 (21.421)
  Dyspnoea score C63D1: number analyzed (Participants) | 53
  Dyspnoea score C63D1 | -1.26 (20.616)
  Dyspnoea score C67D1: number analyzed (Participants) | 46
  Dyspnoea score C67D1 | -3.62 (23.530)
  Dyspnoea score C71D1: number analyzed (Participants) | 43
  Dyspnoea score C71D1 | -3.88 (22.066)
  Dyspnoea score C75D1: number analyzed (Participants) | 24
  Dyspnoea score C75D1 | 0.00 (27.800)
  Dyspnoea score C79D1: number analyzed (Participants) | 20
  Dyspnoea score C79D1 | 1.67 (25.301)
  Dyspnoea score C83D1: number analyzed (Participants) | 8
  Dyspnoea score C83D1 | 12.50 (17.252)
  Dyspnoea score C87D1: number analyzed (Participants) | 2
  Dyspnoea score C87D1 | 50.00 (23.617)
  Dyspnoea score C91D1: number analyzed (Participants) | 1
  Dyspnoea score C91D1 | 66.70
  Dyspnoea score Discontinuation visit: number analyzed (Participants) | 444
  Dyspnoea score Discontinuation visit | 8.71 (29.191)
  Insomnia score Baseline: number analyzed (Participants) | 961
  Insomnia score Baseline | 27.26 (30.907)
  Insomnia score C2D1: number analyzed (Participants) | 812
  Insomnia score C2D1 | -1.35 (28.522)
  Insomnia score C3D1: number analyzed (Participants) | 711
  Insomnia score C3D1 | -1.59 (29.084)
  Insomnia score C4D1: number analyzed (Participants) | 527
  Insomnia score C4D1 | -2.09 (30.102)
  Insomnia score C7D1: number analyzed (Participants) | 349
  Insomnia score C7D1 | -5.92 (31.614)
  Insomnia score C10D1: number analyzed (Participants) | 275
  Insomnia score C10D1 | -5.70 (28.263)
  Insomnia score C13D1: number analyzed (Participants) | 224
  Insomnia score C13D1 | -3.87 (30.033)
  Insomnia score C16D1: number analyzed (Participants) | 189
  Insomnia score C16D1 | -6.88 (33.594)
  Insomnia score C19D1: number analyzed (Participants) | 161
  Insomnia score C19D1 | -6.62 (28.337)
  Insomnia score C23D1: number analyzed (Participants) | 130
  Insomnia score C23D1 | -5.64 (29.969)
  Insomnia score C27D1: number analyzed (Participants) | 122
  Insomnia score C27D1 | -6.28 (29.791)
  Insomnia score C31D1: number analyzed (Participants) | 109
  Insomnia score C31D1 | -12.54 (30.360)
  Insomnia score C35D1: number analyzed (Participants) | 103
  Insomnia score C35D1 | -9.39 (33.797)
  Insomnia score C39D1: number analyzed (Participants) | 91
  Insomnia score C39D1 | -10.26 (33.217)
  Insomnia score C43D1: number analyzed (Participants) | 76
  Insomnia score C43D1 | -4.83 (34.298)
  Insomnia score C47D1: number analyzed (Participants) | 73
  Insomnia score C47D1 | -4.57 (31.091)
  Insomnia score C51D1: number analyzed (Participants) | 70
  Insomnia score C51D1 | -4.28 (28.901)
  Insomnia score C55D1: number analyzed (Participants) | 56
  Insomnia score C55D1 | -2.38 (33.548)
  Insomnia score C59D1: number analyzed (Participants) | 54
  Insomnia score C59D1 | -4.94 (27.784)
  Insomnia score C63D1: number analyzed (Participants) | 53
  Insomnia score C63D1 | -1.89 (29.540)
  Insomnia score C67D1: number analyzed (Participants) | 46
  Insomnia score C67D1 | -4.35 (31.901)
  Insomnia score C71D1: number analyzed (Participants) | 43
  Insomnia score C71D1 | -9.30 (31.972)
  Insomnia score C75D1: number analyzed (Participants) | 24
  Insomnia score C75D1 | -6.95 (29.451)
  Insomnia score C79D1: number analyzed (Participants) | 20
  Insomnia score C79D1 | -6.95 (29.451)
  Insomnia score C83D1: number analyzed (Participants) | 8
  Insomnia score C83D1 | -16.69 (35.646)
  Insomnia score C87D1: number analyzed (Participants) | 2
  Insomnia score C87D1 | -0.05 (47.164)
  Insomnia score C91D1: number analyzed (Participants) | 1
  Insomnia score C91D1 | 33.30
  Insomnia score Discontinuation visit: number analyzed (Participants) | 442
  Insomnia score Discontinuation visit | 8.07 (33.114)
  Appetite Loss score Baseline: number analyzed (Participants) | 960
  Appetite Loss score Baseline | 21.21 (30.066)
  Appetite Loss score C2D1: number analyzed (Participants) | 811
  Appetite Loss score C2D1 | 7.36 (27.805)
  Appetite Loss score C3D1: number analyzed (Participants) | 710
  Appetite Loss score C3D1 | 6.15 (26.405)
  Appetite Loss score C4D1: number analyzed (Participants) | 525
  Appetite Loss score C4D1 | 1.97 (28.206)
  Appetite Loss score C7D1: number analyzed (Participants) | 350
  Appetite Loss score C7D1 | -1.14 (29.837)
  Appetite Loss score C10D1: number analyzed (Participants) | 277
  Appetite Loss score C10D1 | -2.89 (26.152)
  Appetite Loss score C13D1: number analyzed (Participants) | 224
  Appetite Loss score C13D1 | -3.72 (27.719)
  Appetite Loss score C16D1: number analyzed (Participants) | 189
  Appetite Loss score C16D1 | -4.94 (26.392)
  Appetite Loss score C19D1: number analyzed (Participants) | 161
  Appetite Loss score C19D1 | -3.73 (23.565)
  Appetite Loss score C23D1: number analyzed (Participants) | 130
  Appetite Loss score C23D1 | -1.02 (24.532)
  Appetite Loss score C27D1: number analyzed (Participants) | 122
  Appetite Loss score C27D1 | -3.28 (25.136)
  Appetite Loss score C31D1: number analyzed (Participants) | 109
  Appetite Loss score C31D1 | -5.20 (23.643)
  Appetite Loss score C35D1: number analyzed (Participants) | 103
  Appetite Loss score C35D1 | -7.77 (28.847)
  Appetite Loss score C39D1: number analyzed (Participants) | 91
  Appetite Loss score C39D1 | -6.96 (26.064)
  Appetite Loss score C43D1: number analyzed (Participants) | 76
  Appetite Loss score C43D1 | -5.26 (22.473)
  Appetite Loss score C47D1: number analyzed (Participants) | 74
  Appetite Loss score C47D1 | -3.15 (23.515)
  Appetite Loss score C51D1: number analyzed (Participants) | 70
  Appetite Loss score C51D1 | -4.29 (21.919)
  Appetite Loss score C55D1: number analyzed (Participants) | 56
  Appetite Loss score C55D1 | -4.16 (27.749)
  Appetite Loss score C59D1: number analyzed (Participants) | 53
  Appetite Loss score C59D1 | -6.92 (23.892)
  Appetite Loss score C63D1: number analyzed (Participants) | 53
  Appetite Loss score C63D1 | -4.40 (25.347)
  Appetite Loss score C67D1: number analyzed (Participants) | 46
  Appetite Loss score C67D1 | -7.24 (19.765)
  Appetite Loss score C71D1: number analyzed (Participants) | 43
  Appetite Loss score C71D1 | -3.10 (20.328)
  Appetite Loss score C75D1: number analyzed (Participants) | 24
  Appetite Loss score C75D1 | -1.39 (6.797)
  Appetite Loss score C79D1: number analyzed (Participants) | 20
  Appetite Loss score C79D1 | -3.34 (23.929)
  Appetite Loss score C83D1: number analyzed (Participants) | 8
  Appetite Loss score C83D1 | 0.03 (35.639)
  Appetite Loss score C87D1: number analyzed (Participants) | 2
  Appetite Loss score C87D1 | 16.65 (23.547)
  Appetite Loss score C91D1: number analyzed (Participants) | 1
  Appetite Loss score C91D1 | 33.30
  Appetite Loss score Discontinuation visit: number analyzed (Participants) | 445
  Appetite Loss score Discontinuation visit | 14.68 (32.487)
  Constipation score Baseline: number analyzed (Participants) | 962
  Constipation score Baseline | 24.98 (31.584)
  Constipation score C2D1: number analyzed (Participants) | 811
  Constipation score C2D1 | 0.74 (26.700)
  Constipation score C3D1: number analyzed (Participants) | 709
  Constipation score C3D1 | -1.41 (29.876)
  Constipation score C4D1: number analyzed (Participants) | 526
  Constipation score C4D1 | -3.48 (27.560)
  Constipation score C7D1: number analyzed (Participants) | 349
  Constipation score C7D1 | -3.91 (29.908)
  Constipation score C10D1: number analyzed (Participants) | 276
  Constipation score C10D1 | -4.95 (29.467)
  Constipation score C13D1: number analyzed (Participants) | 224
  Constipation score C13D1 | -6.40 (30.010)
  Constipation score C16D1: number analyzed (Participants) | 189
  Constipation score C16D1 | -7.05 (28.513)
  Constipation score C19D1: number analyzed (Participants) | 161
  Constipation score C19D1 | -5.38 (25.523)
  Constipation score C23D1: number analyzed (Participants) | 130
  Constipation score C23D1 | -5.64 (26.619)
  Constipation score C27D1: number analyzed (Participants) | 122
  Constipation score C27D1 | -6.01 (29.384)
  Constipation score C31D1: number analyzed (Participants) | 109
  Constipation score C31D1 | -12.53 (27.131)
  Constipation score C35D1: number analyzed (Participants) | 103
  Constipation score C35D1 | -12.30 (28.388)
  Constipation score C39D1: number analyzed (Participants) | 91
  Constipation score C39D1 | -10.25 (29.267)
  Constipation score C43D1: number analyzed (Participants) | 76
  Constipation score C43D1 | -8.77 (27.953)
  Constipation score C47D1: number analyzed (Participants) | 74
  Constipation score C47D1 | -9.46 (27.868)
  Constipation score C51D1: number analyzed (Participants) | 70
  Constipation score C51D1 | -9.52 (30.108)
  Constipation score C55D1: number analyzed (Participants) | 56
  Constipation score C55D1 | -8.33 (25.624)
  Constipation score C59D1: number analyzed (Participants) | 54
  Constipation score C59D1 | -9.87 (22.079)
  Constipation score C63D1: number analyzed (Participants) | 53
  Constipation score C63D1 | -9.43 (22.052)
  Constipation score C67D1: number analyzed (Participants) | 46
  Constipation score C67D1 | -8.69 (20.408)
  Constipation score C71D1: number analyzed (Participants) | 43
  Constipation score C71D1 | -8.52 (23.112)
  Constipation score C75D1: number analyzed (Participants) | 24
  Constipation score C75D1 | -4.16 (14.933)
  Constipation score C79D1: number analyzed (Participants) | 20
  Constipation score C79D1 | -8.33 (30.334)
  Constipation score C83D1: number analyzed (Participants) | 8
  Constipation score C83D1 | -12.49 (17.234)
  Constipation score C87D1: number analyzed (Participants) | 2
  Constipation score C87D1 | 0.00 (0.00)
  Constipation score C91D1: number analyzed (Participants) | 1
  Constipation score C91D1 | 0.00
  Constipation score Discontinuation visit: number analyzed (Participants) | 444
  Constipation score Discontinuation visit | 4.13 (33.230)
  Diarrhoea score Baseline: number analyzed (Participants) | 960
  Diarrhoea score Baseline | 6.84 (16.552)
  Diarrhoea score C2D1: number analyzed (Participants) | 811
  Diarrhoea score C2D1 | 1.23 (18.840)
  Diarrhoea score C3D1: number analyzed (Participants) | 705
  Diarrhoea score C3D1 | 0.33 (19.495)
  Diarrhoea score C4D1: number analyzed (Participants) | 523
  Diarrhoea score C4D1 | -0.32 (18.847)
  Diarrhoea score C7D1: number analyzed (Participants) | 348
  Diarrhoea score C7D1 | 0.38 (18.060)
  Diarrhoea score C10D1: number analyzed (Participants) | 276
  Diarrhoea score C10D1 | 1.57 (21.110)
  Diarrhoea score C13D1: number analyzed (Participants) | 221
  Diarrhoea score C13D1 | 1.81 (20.267)
  Diarrhoea score C16D1: number analyzed (Participants) | 188
  Diarrhoea score C16D1 | 0.71 (15.774)
  Diarrhoea score C19D1: number analyzed (Participants) | 161
  Diarrhoea score C19D1 | 1.45 (19.838)
  Diarrhoea score C23D1: number analyzed (Participants) | 131
  Diarrhoea score C23D1 | -0.25 (18.251)
  Diarrhoea score C27D1: number analyzed (Participants) | 122
  Diarrhoea score C27D1 | -1.37 (15.677)
  Diarrhoea score C31D1: number analyzed (Participants) | 109
  Diarrhoea score C31D1 | -0.31 (15.374)
  Diarrhoea score C35D1: number analyzed (Participants) | 103
  Diarrhoea score C35D1 | 1.29 (19.755)
  Diarrhoea score C39D1: number analyzed (Participants) | 91
  Diarrhoea score C39D1 | -2.56 (14.252)
  Diarrhoea score C43D1: number analyzed (Participants) | 76
  Diarrhoea score C43D1 | -1.31 (12.684)
  Diarrhoea score C47D1: number analyzed (Participants) | 74
  Diarrhoea score C47D1 | -2.25 (15.915)
  Diarrhoea score C51D1: number analyzed (Participants) | 71
  Diarrhoea score C51D1 | -1.41 (15.356)
  Diarrhoea score C55D1: number analyzed (Participants) | 56
  Diarrhoea score C55D1 | -1.19 (10.933)
  Diarrhoea score C59D1: number analyzed (Participants) | 54
  Diarrhoea score C59D1 | -1.85 (13.595)
  Diarrhoea score C63D1: number analyzed (Participants) | 53
  Diarrhoea score C63D1 | -1.26 (11.240)
  Diarrhoea score C67D1: number analyzed (Participants) | 46
  Diarrhoea score C67D1 | -1.45 (13.964)
  Diarrhoea score C71D1: number analyzed (Participants) | 43
  Diarrhoea score C71D1 | -2.32 (13.390)
  Diarrhoea score C75D1: number analyzed (Participants) | 25
  Diarrhoea score C75D1 | -1.33 (15.138)
  Diarrhoea score C79D1: number analyzed (Participants) | 20
  Diarrhoea score C79D1 | -3.33 (14.892)
  Diarrhoea score C83D1: number analyzed (Participants) | 8
  Diarrhoea score C83D1 | 4.16 (21.341)
  Diarrhoea score C87D1: number analyzed (Participants) | 2
  Diarrhoea score C87D1 | 0.00 (0.00)
  Diarrhoea score C91D1: number analyzed (Participants) | 1
  Diarrhoea score C91D1 | 0.00
  Diarrhoea score Discontinuation visit: number analyzed (Participants) | 440
  Diarrhoea score Discontinuation visit | 0.30 (22.379)
  Financial difficulties score Baseline: number analyzed (Participants) | 959
  Financial difficulties score Baseline | 17.34 (27.147)
  Financial difficulties score C2D1: number analyzed (Participants) | 807
  Financial difficulties score C2D1 | -1.86 (21.216)
  Financial difficulties score C3D1: number analyzed (Participants) | 702
  Financial difficulties score C3D1 | -1.42 (22.408)
  Financial difficulties score C4D1: number analyzed (Participants) | 521
  Financial difficulties score C4D1 | -1.54 (22.497)
  Financial difficulties score C7D1: number analyzed (Participants) | 346
  Financial difficulties score C7D1 | -4.14 (24.057)
  Financial difficulties score C10D1: number analyzed (Participants) | 275
  Financial difficulties score C10D1 | -3.88 (24.021)
  Financial difficulties score C13D1: number analyzed (Participants) | 222
  Financial difficulties score C13D1 | -4.06 (22.615)
  Financial difficulties score C16D1: number analyzed (Participants) | 188
  Financial difficulties score C16D1 | -2.84 (25.172)
  Financial difficulties score C19D1: number analyzed (Participants) | 161
  Financial difficulties score C19D1 | -4.14 (26.023)
  Financial difficulties score C23D1: number analyzed (Participants) | 131
  Financial difficulties score C23D1 | -5.35 (24.042)
  Financial difficulties score C27D1: number analyzed (Participants) | 122
  Financial difficulties score C27D1 | -5.19 (23.867)
  Financial difficulties score C31D1: number analyzed (Participants) | 109
  Financial difficulties score C31D1 | -9.48 (26.489)
  Financial difficulties score C35D1: number analyzed (Participants) | 101
  Financial difficulties score C35D1 | -3.96 (25.517)
  Financial difficulties score C39D1: number analyzed (Participants) | 91
  Financial difficulties score C39D1 | -4.76 (25.615)
  Financial difficulties score C43D1: number analyzed (Participants) | 76
  Financial difficulties score C43D1 | -2.63 (22.942)
  Financial difficulties score C47D1: number analyzed (Participants) | 74
  Financial difficulties score C47D1 | -0.90 (25.869)
  Financial difficulties score C51D1: number analyzed (Participants) | 71
  Financial difficulties score C51D1 | -5.63 (25.191)
  Financial difficulties score C55D1: number analyzed (Participants) | 56
  Financial difficulties score C55D1 | -4.76 (26.541)
  Financial difficulties score C59D1: number analyzed (Participants) | 54
  Financial difficulties score C59D1 | -6.79 (24.551)
  Financial difficulties score C63D1: number analyzed (Participants) | 53
  Financial difficulties score C63D1 | -6.92 (22.984)
  Financial difficulties score C67D1: number analyzed (Participants) | 46
  Financial difficulties score C67D1 | -6.52 (24.963)
  Financial difficulties score C71D1: number analyzed (Participants) | 43
  Financial difficulties score C71D1 | -6.98 (17.154)
  Financial difficulties score C75D1: number analyzed (Participants) | 25
  Financial difficulties score C75D1 | -14.68 (23.740)
  Financial difficulties score C79D1: number analyzed (Participants) | 20
  Financial difficulties score C79D1 | -1.68 (20.157)
  Financial difficulties score C83D1: number analyzed (Participants) | 8
  Financial difficulties score C83D1 | -4.18 (33.028)
  Financial difficulties score C87D1: number analyzed (Participants) | 2
  Financial difficulties score C87D1 | -16.70 (23.617)
  Financial difficulties score C91D1: number analyzed (Participants) | 1
  Financial difficulties score C91D1 | 0.00
  Financial difficulties score Discontinuation visit: number analyzed (Participants) | 442
  Financial difficulties score Discontinuation visit | 2.41 (27.481)
  Global health status Baseline: number analyzed (Participants) | 962
  Global health status Baseline | 59.01 (22.821)
  Global health status C2D1: number analyzed (Participants) | 813
  Global health status C2D1 | -1.48 (19.541)
  Global health status C3D1: number analyzed (Participants) | 708
  Global health status C3D1 | -0.27 (19.770)
  Global health status C4D1: number analyzed (Participants) | 526
  Global health status C4D1 | 0.82 (20.587)
  Global health status C7D1: number analyzed (Participants) | 350
  Global health status C7D1 | 3.64 (20.564)
  Global health status C10D1: number analyzed (Participants) | 278
  Global health status C10D1 | 3.63 (19.943)
  Global health status C13D1: number analyzed (Participants) | 222
  Global health status C13D1 | 6.01 (19.679)
  Global health status C16D1: number analyzed (Participants) | 188
  Global health status C16D1 | 5.76 (21.404)
  Global health status C19D1: number analyzed (Participants) | 162
  Global health status C19D1 | 4.88 (20.838)
  Global health status C23D1: number analyzed (Participants) | 131
  Global health status C23D1 | 5.21 (21.759)
  Global health status C27D1: number analyzed (Participants) | 122
  Global health status C27D1 | 6.22 (24.016)
  Global health status C31D1: number analyzed (Participants) | 109
  Global health status C31D1 | 8.10 (22.827)
  Global health status C35D1: number analyzed (Participants) | 103
  Global health status C35D1 | 11.17 (22.555)
  Global health status C39D1: number analyzed (Participants) | 91
  Global health status C39D1 | 8.52 (23.857)
  Global health status C43D1: number analyzed (Participants) | 76
  Global health status C43D1 | 8.56 (22.846)
  Global health status C47D1: number analyzed (Participants) | 74
  Global health status C47D1 | 5.30 (24.608)
  Global health status C51D1: number analyzed (Participants) | 71
  Global health status C51D1 | 7.51 (20.985)
  Global health status C55D1: number analyzed (Participants) | 56
  Global health status C55D1 | 8.49 (20.309)
  Global health status C59D1: number analyzed (Participants) | 54
  Global health status C59D1 | 9.57 (18.900)
  Global health status C63D1: number analyzed (Participants) | 53
  Global health status C63D1 | 8.34 (19.604)
  Global health status C67D1: number analyzed (Participants) | 46
  Global health status C67D1 | 7.43 (22.369)
  Global health status C71D1: number analyzed (Participants) | 43
  Global health status C71D1 | 9.30 (21.904)
  Global health status C75D1: number analyzed (Participants) | 25
  Global health status C75D1 | 10.67 (19.301)
  Global health status C79D1: number analyzed (Participants) | 20
  Global health status C79D1 | 10.43 (16.196)
  Global health status C83D1: number analyzed (Participants) | 8
  Global health status C83D1 | 10.44 (15.292)
  Global health status C87D1: number analyzed (Participants) | 2
  Global health status C87D1 | 4.20 (17.678)
  Global health status C91D1: number analyzed (Participants) | 1
  Global health status C91D1 | -8.30
  Global health status Discontinuation visit: number analyzed (Participants) | 444
  Global health status Discontinuation visit | -10.94 (27.334)

12. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQoL) Group 5-Dimension 5-Level (EQ-5D-5L) Self Report Questionnaire Health Utility Score
Description: The EuroQol 5-Dimension Questionnaire (EQ-5D-5L) is a self-report health status questionnaire that consists of 6 questions used to calculate a health utility score for use in health economic analysis. There are two components to the EuroQol EQ-5D: 1) five health dimensions that assess mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; 2) a visual analogue scale (VAS) that measures health state. There are 5 response levels for each dimension (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems) with the highest level representing the worst outcome. The VAS is scored on a scale from 0 to 100, with 0 representing the worst imaginable health and 100 representing the best imaginable health.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Atezolizumab
Number analyzed (Participants) | 960
Score on a scale
  Mobility Baseline: number analyzed (Participants) | 958
  Mobility Baseline | 1.9 (1.03)
  Mobility C2D1: number analyzed (Participants) | 809
  Mobility C2D1 | 0.1 (0.81)
  Mobility C3D1: number analyzed (Participants) | 705
  Mobility C3D1 | 0.2 (0.90)
  Mobility C4D1: number analyzed (Participants) | 527
  Mobility C4D1 | 0.1 (0.88)
  Mobility C7D1: number analyzed (Participants) | 344
  Mobility C7D1 | 0.0 (0.93)
  Mobility C10D1: number analyzed (Participants) | 272
  Mobility C10D1 | -0.1 (0.90)
  Mobility C13D1: number analyzed (Participants) | 225
  Mobility C13D1 | -0.1 (0.80)
  Mobility C16D1: number analyzed (Participants) | 189
  Mobility C16D1 | -0.2 (0.91)
  Mobility C19D1: number analyzed (Participants) | 162
  Mobility C19D1 | -0.1 (0.92)
  Mobility C23D1: number analyzed (Participants) | 131
  Mobility C23D1 | -0.1 (0.91)
  Mobility C27D1: number analyzed (Participants) | 121
  Mobility C27D1 | -0.2 (0.84)
  Mobility C31D1: number analyzed (Participants) | 110
  Mobility C31D1 | -0.2 (0.88)
  Mobility C35D1: number analyzed (Participants) | 102
  Mobility C35D1 | -0.1 (1.05)
  Mobility C39D1: number analyzed (Participants) | 93
  Mobility C39D1 | -0.2 (0.92)
  Mobility C43D1: number analyzed (Participants) | 76
  Mobility C43D1 | -0.2 (1.04)
  Mobility C47D1: number analyzed (Participants) | 73
  Mobility C47D1 | -0.2 (0.84)
  Mobility C51D1: number analyzed (Participants) | 72
  Mobility C51D1 | -0.3 (0.89)
  Mobility C55D1: number analyzed (Participants) | 55
  Mobility C55D1 | -0.1 (0.79)
  Mobility C59D1: number analyzed (Participants) | 54
  Mobility C59D1 | -0.2 (0.99)
  Mobility C63D1: number analyzed (Participants) | 52
  Mobility C63D1 | -0.2 (1.00)
  Mobility C67D1: number analyzed (Participants) | 45
  Mobility C67D1 | -0.2 (0.93)
  Mobility C71D1: number analyzed (Participants) | 41
  Mobility C71D1 | -0.1 (0.85)
  Mobility C75D1: number analyzed (Participants) | 25
  Mobility C75D1 | -0.1 (0.67)
  Mobility C79D1: number analyzed (Participants) | 20
  Mobility C79D1 | 0.0 (0.97)
  Mobility C83D1: number analyzed (Participants) | 8
  Mobility C83D1 | -0.1 (0.83)
  Mobility C87D1: number analyzed (Participants) | 2
  Mobility C87D1 | 1.0 (1.41)
  Mobility C91D1: number analyzed (Participants) | 1
  Mobility C91D1 | 2.0
  Mobility Discontinuation visit: number analyzed (Participants) | 439
  Mobility Discontinuation visit | 0.5 (1.19)
  Self-Care Baseline: number analyzed (Participants) | 959
  Self-Care Baseline | 1.4 (0.81)
  Self-Care C2D1: number analyzed (Participants) | 812
  Self-Care C2D1 | 0.1 (0.72)
  Self-Care C3D1: number analyzed (Participants) | 706
  Self-Care C3D1 | 0.2 (0.77)
  Self-Care C4D1: number analyzed (Participants) | 526
  Self-Care C4D1 | 0.1 (0.69)
  Self-Care C7D1: number analyzed (Participants) | 344
  Self-Care C7D1 | 0.0 (0.72)
  Self-Care C10D1: number analyzed (Participants) | 273
  Self-Care C10D1 | 0.0 (0.68)
  Self-Care C13D1: number analyzed (Participants) | 224
  Self-Care C13D1 | 0.0 (0.62)
  Self-Care C16D1: number analyzed (Participants) | 189
  Self-Care C16D1 | -0.1 (0.57)
  Self-Care C19D1: number analyzed (Participants) | 162
  Self-Care C19D1 | 0.0 (0.68)
  Self-Care C23D1: number analyzed (Participants) | 131
  Self-Care C23D1 | 0.0 (0.67)
  Self-Care C27D1: number analyzed (Participants) | 121
  Self-Care C27D1 | 0.0 (0.63)
  Self-Care C31D1: number analyzed (Participants) | 110
  Self-Care C31D1 | -0.1 (0.62)
  Self-Care C35D1: number analyzed (Participants) | 102
  Self-Care C35D1 | -0.1 (0.69)
  Self-Care C39D1: number analyzed (Participants) | 92
  Self-Care C39D1 | -0.1 (0.69)
  Self-Care C43D1: number analyzed (Participants) | 75
  Self-Care C43D1 | -0.1 (0.83)
  Self-Care C47D1: number analyzed (Participants) | 74
  Self-Care C47D1 | -0.1 (0.72)
  Self-Care C51D1: number analyzed (Participants) | 73
  Self-Care C51D1 | -0.1 (0.84)
  Self-Care C55D1: number analyzed (Participants) | 56
  Self-Care C55D1 | -0.1 (0.66)
  Self-Care C59D1: number analyzed (Participants) | 55
  Self-Care C59D1 | -0.1 (0.82)
  Self-Care C63D1: number analyzed (Participants) | 53
  Self-Care C63D1 | -0.1 (0.76)
  Self-Care C67D1: number analyzed (Participants) | 46
  Self-Care C67D1 | -0.1 (0.75)
  Self-Care C71D1: number analyzed (Participants) | 42
  Self-Care C71D1 | 0.0 (0.60)
  Self-Care C75D1: number analyzed (Participants) | 25
  Self-Care C75D1 | 0.0 (0.20)
  Self-Care C79D1: number analyzed (Participants) | 20
  Self-Care C79D1 | 0.1 (0.45)
  Self-Care C83D1: number analyzed (Participants) | 8
  Self-Care C83D1 | -0.3 (0.46)
  Self-Care C87D1: number analyzed (Participants) | 2
  Self-Care C87D1 | 0.0 (0.00)
  Self-Care C91D1: number analyzed (Participants) | 1
  Self-Care C91D1 | 1.0
  Self-Care Discontinuation visit: number analyzed (Participants) | 438
  Self-Care Discontinuation visit | 0.4 (1.04)
  Usual Activities Baseline: number analyzed (Participants) | 959
  Usual Activities Baseline | 2.0 (1.08)
  Usual Activities C2D1: number analyzed (Participants) | 811
  Usual Activities C2D1 | 0.2 (0.92)
  Usual Activities C3D1: number analyzed (Participants) | 706
  Usual Activities C3D1 | 0.2 (0.99)
  Usual Activities C4D1: number analyzed (Participants) | 526
  Usual Activities C4D1 | 0.1 (0.90)
  Usual Activities C7D1: number analyzed (Participants) | 345
  Usual Activities C7D1 | 0.0 (0.93)
  Usual Activities C10D1: number analyzed (Participants) | 273
  Usual Activities C10D1 | -0.1 (0.92)
  Usual Activities C13D1: number analyzed (Participants) | 225
  Usual Activities C13D1 | -0.2 (0.86)
  Usual Activities C16D1: number analyzed (Participants) | 189
  Usual Activities C16D1 | -0.1 (1.04)
  Usual Activities C19D1: number analyzed (Participants) | 163
  Usual Activities C19D1 | 0.0 (0.98)
  Usual Activities C23D1: number analyzed (Participants) | 132
  Usual Activities C23D1 | -0.1 (0.93)
  Usual Activities C27D1: number analyzed (Participants) | 122
  Usual Activities C27D1 | -0.2 (0.92)
  Usual Activities C31D1: number analyzed (Participants) | 111
  Usual Activities C31D1 | -0.3 (0.96)
  Usual Activities C35D1: number analyzed (Participants) | 102
  Usual Activities C35D1 | -0.2 (1.10)
  Usual Activities C39D1: number analyzed (Participants) | 93
  Usual Activities C39D1 | -0.2 (0.96)
  Usual Activities C43D1: number analyzed (Participants) | 76
  Usual Activities C43D1 | -0.1 (0.93)
  Usual Activities C47D1: number analyzed (Participants) | 74
  Usual Activities C47D1 | -0.2 (0.86)
  Usual Activities C51D1: number analyzed (Participants) | 73
  Usual Activities C51D1 | -0.3 (0.91)
  Usual Activities C55D1: number analyzed (Participants) | 56
  Usual Activities C55D1 | -0.2 (0.91)
  Usual Activities C59D1: number analyzed (Participants) | 55
  Usual Activities C59D1 | -0.3 (0.95)
  Usual Activities C63D1: number analyzed (Participants) | 53
  Usual Activities C63D1 | -0.2 (0.85)
  Usual Activities C67D1: number analyzed (Participants) | 46
  Usual Activities C67D1 | -0.3 (0.80)
  Usual Activities C71D1: number analyzed (Participants) | 42
  Usual Activities C71D1 | -0.2 (0.68)
  Usual Activities C75D1: number analyzed (Participants) | 25
  Usual Activities C75D1 | -0.1 (0.49)
  Usual Activities C79D1: number analyzed (Participants) | 20
  Usual Activities C79D1 | 0.0 (0.65)
  Usual Activities C83D1: number analyzed (Participants) | 8
  Usual Activities C83D1 | 0.1 (0.64)
  Usual Activities C87D1: number analyzed (Participants) | 2
  Usual Activities C87D1 | 0.0 (0.00)
  Usual Activities C91D1: number analyzed (Participants) | 1
  Usual Activities C91D1 | 0.0
  Usual Activities Discontinuation visit: number analyzed (Participants) | 438
  Usual Activities Discontinuation visit | 0.6 (1.23)
  Pain/Discomfort Baseline: number analyzed (Participants) | 959
  Pain/Discomfort Baseline | 2.3 (1.08)
  Pain/Discomfort C2D1: number analyzed (Participants) | 810
  Pain/Discomfort C2D1 | 0.0 (0.82)
  Pain/Discomfort C3D1: number analyzed (Participants) | 706
  Pain/Discomfort C3D1 | 0.1 (0.98)
  Pain/Discomfort C4D1: number analyzed (Participants) | 524
  Pain/Discomfort C4D1 | 0.0 (0.94)
  Pain/Discomfort C7D1: number analyzed (Participants) | 344
  Pain/Discomfort C7D1 | 0.0 (1.04)
  Pain/Discomfort C10D1: number analyzed (Participants) | 274
  Pain/Discomfort C10D1 | -0.2 (0.96)
  Pain/Discomfort C13D1: number analyzed (Participants) | 226
  Pain/Discomfort C13D1 | -0.2 (0.96)
  Pain/Discomfort C16D1: number analyzed (Participants) | 190
  Pain/Discomfort C16D1 | -0.3 (1.02)
  Pain/Discomfort C19D1: number analyzed (Participants) | 163
  Pain/Discomfort C19D1 | -0.2 (1.04)
  Pain/Discomfort C23D1: number analyzed (Participants) | 132
  Pain/Discomfort C23D1 | -0.2 (1.04)
  Pain/Discomfort C27D1: number analyzed (Participants) | 122
  Pain/Discomfort C27D1 | -0.3 (1.03)
  Pain/Discomfort C31D1: number analyzed (Participants) | 11
  Pain/Discomfort C31D1 | -0.3 (0.96)
  Pain/Discomfort C35D1: number analyzed (Participants) | 103
  Pain/Discomfort C35D1 | -0.3 (1.15)
  Pain/Discomfort C39D1: number analyzed (Participants) | 93
  Pain/Discomfort C39D1 | -0.4 (1.05)
  Pain/Discomfort C43D1: number analyzed (Participants) | 76
  Pain/Discomfort C43D1 | -0.4 (0.98)
  Pain/Discomfort C47D1: number analyzed (Participants) | 74
  Pain/Discomfort C47D1 | -0.4 (1.03)
  Pain/Discomfort C51D1: number analyzed (Participants) | 73
  Pain/Discomfort C51D1 | -0.3 (1.07)
  Pain/Discomfort C55D1: number analyzed (Participants) | 56
  Pain/Discomfort C55D1 | -0.4 (1.00)
  Pain/Discomfort C59D1: number analyzed (Participants) | 55
  Pain/Discomfort C59D1 | -0.4 (1.05)
  Pain/Discomfort C63D1: number analyzed (Participants) | 53
  Pain/Discomfort C63D1 | -0.3 (1.04)
  Pain/Discomfort C67D1: number analyzed (Participants) | 46
  Pain/Discomfort C67D1 | -0.2 (1.20)
  Pain/Discomfort C71D1: number analyzed (Participants) | 42
  Pain/Discomfort C71D1 | -0.2 (1.09)
  Pain/Discomfort C75D1: number analyzed (Participants) | 25
  Pain/Discomfort C75D1 | -0.3 (1.11)
  Pain/Discomfort C79D1: number analyzed (Participants) | 20
  Pain/Discomfort C79D1 | -0.3 (1.02)
  Pain/Discomfort C83D1: number analyzed (Participants) | 8
  Pain/Discomfort C83D1 | 0.0 (0.93)
  Pain/Discomfort C87D1: number analyzed (Participants) | 2
  Pain/Discomfort C87D1 | -1.0 (0.00)
  Pain/Discomfort C91D1: number analyzed (Participants) | 1
  Pain/Discomfort C91D1 | 0.0
  Pain/Discomfort Discontinuation visit: number analyzed (Participants) | 439
  Pain/Discomfort Discontinuation visit | 0.3 (1.18)
  Anxiety/Depression Baseline | 1.7 (0.87)
  Anxiety/Depression C2D1: number analyzed (Participants) | 812
  Anxiety/Depression C2D1 | 0.0 (0.75)
  Anxiety/Depression C3D1: number analyzed (Participants) | 707
  Anxiety/Depression C3D1 | 0.0 (0.81)
  Anxiety/Depression C4D1: number analyzed (Participants) | 526
  Anxiety/Depression C4D1 | 0.0 (0.87)
  Anxiety/Depression C7D1: number analyzed (Participants) | 344
  Anxiety/Depression C7D1 | -0.1 (0.81)
  Anxiety/Depression C10D1: number analyzed (Participants) | 272
  Anxiety/Depression C10D1 | -0.2 (0.74)
  Anxiety/Depression C13D1: number analyzed (Participants) | 224
  Anxiety/Depression C13D1 | -0.2 (0.78)
  Anxiety/Depression C16D1: number analyzed (Participants) | 190
  Anxiety/Depression C16D1 | -0.2 (0.78)
  Anxiety/Depression C19D1: number analyzed (Participants) | 163
  Anxiety/Depression C19D1 | -0.1 (0.78)
  Anxiety/Depression C23D1: number analyzed (Participants) | 132
  Anxiety/Depression C23D1 | -0.1 (0.88)
  Anxiety/Depression C27D1: number analyzed (Participants) | 122
  Anxiety/Depression C27D1 | -0.2 (0.73)
  Anxiety/Depression C31D1: number analyzed (Participants) | 111
  Anxiety/Depression C31D1 | -0.3 (0.75)
  Anxiety/Depression C35D1: number analyzed (Participants) | 102
  Anxiety/Depression C35D1 | -0.3 (0.74)
  Anxiety/Depression C39D1: number analyzed (Participants) | 93
  Anxiety/Depression C39D1 | -0.2 (0.78)
  Anxiety/Depression C43D1: number analyzed (Participants) | 76
  Anxiety/Depression C43D1 | -0.3 (0.80)
  Anxiety/Depression C47D1: number analyzed (Participants) | 74
  Anxiety/Depression C47D1 | -0.3 (0.77)
  Anxiety/Depression C51D1: number analyzed (Participants) | 73
  Anxiety/Depression C51D1 | -0.2 (0.78)
  Anxiety/Depression C55D1: number analyzed (Participants) | 56
  Anxiety/Depression C55D1 | -0.2 (0.73)
  Anxiety/Depression C59D1: number analyzed (Participants) | 55
  Anxiety/Depression C59D1 | -0.1 (0.68)
  Anxiety/Depression C63D1: number analyzed (Participants) | 51
  Anxiety/Depression C63D1 | -0.1 (0.82)
  Anxiety/Depression C67D1: number analyzed (Participants) | 46
  Anxiety/Depression C67D1 | -0.1 (0.76)
  Anxiety/Depression C71D1: number analyzed (Participants) | 42
  Anxiety/Depression C71D1 | -0.1 (0.78)
  Anxiety/Depression C75D1: number analyzed (Participants) | 24
  Anxiety/Depression C75D1 | -0.3 (0.82)
  Anxiety/Depression C79D1: number analyzed (Participants) | 20
  Anxiety/Depression C79D1 | -0.5 (1.00)
  Anxiety/Depression C83D1: number analyzed (Participants) | 8
  Anxiety/Depression C83D1 | -0.4 (0.74)
  Anxiety/Depression C87D1: number analyzed (Participants) | 2
  Anxiety/Depression C87D1 | 0.0 (1.41)
  Anxiety/Depression C91D1: number analyzed (Participants) | 1
  Anxiety/Depression C91D1 | 1.0
  Anxiety/Depression Discontinuation visit: number analyzed (Participants) | 438
  Anxiety/Depression Discontinuation visit | 0.3 (1.03)
  Visual Analog Scale (VAS) Baseline: number analyzed (Participants) | 958
  Visual Analog Scale (VAS) Baseline | 64.7 (20.37)
  VAS C2D1: number analyzed (Participants) | 808
  VAS C2D1 | -0.6 (14.76)
  VAS C3D1: number analyzed (Participants) | 703
  VAS C3D1 | -0.3 (17.21)
  VAS C4D1: number analyzed (Participants) | 528
  VAS C4D1 | 0.3 (18.02)
  VAS C7D1: number analyzed (Participants) | 344
  VAS C7D1 | 3.7 (17.47)
  VAS C10D1: number analyzed (Participants) | 274
  VAS C10D1 | 3.5 (17.88)
  VAS C13D1: number analyzed (Participants) | 222
  VAS C13D1 | 5.8 (17.46)
  VAS C16D1: number analyzed (Participants) | 190
  VAS C16D1 | 6.4 (17.87)
  VAS C19D1: number analyzed (Participants) | 162
  VAS C19D1 | 5.9 (16.49)
  VAS C23D1: number analyzed (Participants) | 132
  VAS C23D1 | 7.7 (17.14)
  VAS C27D1: number analyzed (Participants) | 111
  VAS C27D1 | 8.9 (17.99)
  VAS C31D1: number analyzed (Participants) | 111
  VAS C31D1 | 8.9 (17.99)
  VAS C35D1: number analyzed (Participants) | 103
  VAS C35D1 | 11.0 (19.13)
  VAS C39D1: number analyzed (Participants) | 93
  VAS C39D1 | 9.0 (19.31)
  VAS C43D1: number analyzed (Participants) | 76
  VAS C43D1 | 8.9 (17.59)
  VAS C47D1: number analyzed (Participants) | 75
  VAS C47D1 | 9.0 (16.08)
  VAS C51D1: number analyzed (Participants) | 73
  VAS C51D1 | 7.4 (18.85)
  VAS C55D1: number analyzed (Participants) | 57
  VAS C55D1 | 8.7 (18.10)
  VAS C59D1: number analyzed (Participants) | 55
  VAS C59D1 | 5.3 (16.15)
  VAS C63D1: number analyzed (Participants) | 54
  VAS C63D1 | 8.5 (17.08)
  VAS C67D1: number analyzed (Participants) | 47
  VAS C67D1 | 6.8 (18.89)
  VAS C71D1: number analyzed (Participants) | 42
  VAS C71D1 | 7.7 (18.48)
  VAS C75D1: number analyzed (Participants) | 25
  VAS C75D1 | 8.3 (14.89)
  VAS C79D1: number analyzed (Participants) | 20
  VAS C79D1 | 7.2 (13.47)
  VAS C83D1: number analyzed (Participants) | 8
  VAS C83D1 | 9.0 (10.74)
  VAS C87D1: number analyzed (Participants) | 2
  VAS C87D1 | 7.5 (10.61)
  VAS C91D1: number analyzed (Participants) | 1
  VAS C91D1 | 0.0
  VAS Discontinuation visit: number analyzed (Participants) | 437
  VAS Discontinuation visit | -8.0 (22.60)

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to approximately 6 years)
Description: All-cause mortality is reported for deaths that occurred during the study based on the ITT population, which included all randomized participants regardless of whether the assigned study treatment was received. Serious and other AEs were reported based on the safety population, which included all randomized participants who received any amount of study treatment, regardless of whether a full or partial dose was received. This population was evaluated after the initiation of study treatment.
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 780/1004
Serious Adverse Events (participants affected / at risk) | 380/997
Other Adverse Events (participants affected / at risk) | 888/997
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (N=997)
Urinary tract infection (Infections and infestations) | 59
Urosepsis (Infections and infestations) | 19
Pneumonia (Infections and infestations) | 17
Sepsis (Infections and infestations) | 12
Intestinal obstruction (Gastrointestinal disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 10
Haematuria (Renal and urinary disorders) | 19
Acute kidney injury (Renal and urinary disorders) | 16
Pyrexia (General disorders) | 15
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11
Pyelonephritis (Infections and infestations) | 7
Cellulitis (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 5
Infection (Infections and infestations) | 4
Septic shock (Infections and infestations) | 4
Device related infection (Infections and infestations) | 3
Erysipelas (Infections and infestations) | 3
Lower respiratory tract infection (Infections and infestations) | 3
Postoperative wound infection (Infections and infestations) | 3
Cystitis (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Encephalitis (Infections and infestations) | 2
Endocarditis (Infections and infestations) | 2
Febrile infection (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 2
Scrotal abscess (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 2
Urinary tract infection bacterial (Infections and infestations) | 2
Vascular device infection (Infections and infestations) | 2
Abdominal infection (Infections and infestations) | 1
Abdominal sepsis (Infections and infestations) | 1
Acute hepatitis B (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Candida sepsis (Infections and infestations) | 1
Chlamydial infection (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Infective aneurysm (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Post procedural sepsis (Infections and infestations) | 1
Respiratory moniliasis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Stoma site infection (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Colitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 2
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Renal failure (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 5
Urinary tract obstruction (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 3
Hydronephrosis (Renal and urinary disorders) | 3
Nephritis (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 2
Bladder tamponade (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1
Death (General disorders) | 8
Fatigue (General disorders) | 4
Chest pain (General disorders) | 2
General physical health deterioration (General disorders) | 2
Pain (General disorders) | 2
Asthenia (General disorders) | 1
Complication of device insertion (General disorders) | 1
Hyperpyrexia (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Performance status decreased (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Vascular device occlusion (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Cardiac failure (Cardiac disorders) | 5
Myocardial infarction (Cardiac disorders) | 4
Acute myocardial infarction (Cardiac disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericardial haemorrhage (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Autoimmune hepatitis (Hepatobiliary disorders) | 2
Hepatitis (Hepatobiliary disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 2
Acute hepatic failure (Hepatobiliary disorders) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Hepatic cyst (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Cerebrovascular accident (Nervous system disorders) | 2
Aphasia (Nervous system disorders) | 1
Cerebral atrophy (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Intermittent claudication (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Blood creatinine increased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Myocardial necrosis marker increased (Investigations) | 1
Transaminases increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Device occlusion (Product Issues) | 4
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Scrotal inflammation (Reproductive system and breast disorders) | 1
Spermatocele (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hypophysitis (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Systemic immune activation (Immune system disorders) | 2
Sarcoidosis (Immune system disorders) | 1
Corneal degeneration (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (N=997)
Asthenia (General disorders) | 211
Fatigue (General disorders) | 206
Pyrexia (General disorders) | 156
Oedema peripheral (General disorders) | 64
Diarrhoea (Gastrointestinal disorders) | 166
Constipation (Gastrointestinal disorders) | 145
Nausea (Gastrointestinal disorders) | 130
Vomiting (Gastrointestinal disorders) | 103
Abdominal pain (Gastrointestinal disorders) | 62
Urinary tract infection (Infections and infestations) | 152
Arthralgia (Musculoskeletal and connective tissue disorders) | 132
Back pain (Musculoskeletal and connective tissue disorders) | 120
Pain in extremity (Musculoskeletal and connective tissue disorders) | 64
Decreased appetite (Metabolism and nutrition disorders) | 185
Pruritus (Skin and subcutaneous tissue disorders) | 125
Rash (Skin and subcutaneous tissue disorders) | 72
Blood creatinine increased (Investigations) | 70
Anaemia (Blood and lymphatic system disorders) | 182
Haematuria (Renal and urinary disorders) | 76
Cough (Respiratory, thoracic and mediastinal disorders) | 104
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 72
Hypothyroidism (Endocrine disorders) | 67
Pain (General disorders) | 57
Weight decreased (Investigations) | 50
Headache (Nervous system disorders) | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT02928406/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT02928406/SAP_001.pdf